CLINICAL TRIAL: NCT02531893
Title: Psychological Treatments for Youth With Severe Irritability
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150182; 15-M-0182
Record Dates: First submitted 2015-08-22; First posted 2015-08-25 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-11-19

CONDITIONS: Irritability
Keywords: Interpretation Bias Training; Cognitive Behavioral Therapy; Children; Natural History

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Irritable youth: Participants meet full DMDD criteria for IBT and either full DMDD or one of two core DMDD criteria for CBT.

SUMMARY:
Background:

When children have severe irritability and temper outbursts, they can be so cranky or angry that it leads to problems at home, in school, and with friends. This is called Disruptive Mood Dysregulation Disorder (DMDD) and there have been no psychological treatments developed specifically for children with this problem. Researchers think two forms of therapy, Cognitive Behavioral Therapy (CBT) and Interpretation Bias Training (IBT), might help children with DMDD.

Objective:

To test two whether IBT and CBT can decrease severe irritability in children and youth.

Eligibility:

Children 8-17 years old with DMDD. Their symptoms must have started before age 10.

Design:

Participants will be screened with a review of their symptoms. Parents and participants will answer questions.

Participants can do only one or both of these treatments if they wish. Those who wish to do both will start with IBT.

Participants who do CBT will have 12-16 weekly meetings of research talk therapy. A parent will participate in part of the sessions.

Participants will talk about what makes them irritable and how it affects them. They may be put in situations that might make them annoyed or irritable.

Participants will rate how intense their irritability is. Parents and participants will complete rating scales, questionnaires, and interviews.

Participants will do practice activities at home.

Participants doing IBT will have up to 14 sessions over 10 weeks.

Participants will view 15 faces, one at a time, on a computer. They will choose if the face looks happy or angry on a computer. Sometimes the computer gives feedback. Participants will complete some sessions at the NIH and some at home.

Participants and parents answer questions about their progress.

DETAILED DESCRIPTION:
OBJECTIVE:

This purpose of this protocol is to further the development of two potential non-pharmacologic treatments for youths with chronic, severe and impairing irritability. The first potential treatment is Interpretation Bias Training (IBT), a computer-based training designed to shift emotional judgments of ambiguous faces away from angry, and toward happy, judgments. The first component of this protocol includes a randomized, controlled trial of active IBT in youth with severe irritability. The second potential treatment is a cognitive behavioral therapy (CBT) targeting severe irritability. The goal of this protocol is to conduct a preliminary study using a randomized within-subjects multiple-baseline design to test the efficacy of a new manualized exposure-based CBT with parenting training in the treatment of severe irritability.

Objective 1: Assess the efficacy of Interpretation Bias Training (IBT) in youths with severe irritability, operationalized as those meeting criteria for DSM-5 Disruptive Mood Dysregulation Disorder (DMDD). To accomplish this objective, we will conduct a randomized, controlled trial (RCT) of active IBT in 40 youths with DMDD. Subjects will be randomized to receive four IBT training sessions (active vs. placebo, in a double-blind design) over four days followed by weekly mood ratings for two weeks. Primary outcome measures in this trial will assess changes in irritability using the Affective Reactivity Index (ARI: clinician-rated, parent-rated, and child-rated) and Clinical Global Impressions-Improvement (CGI-I). After completing the RCT, all participants will be offered four open, active IBT sessions, delivered on the same schedule as in the RCT and using the same primary outcome measures.

Objective 2: Test the efficacy of a new manualized CBT for severe, impairing irritability in youth and adapt the in-person manual to being a hybrid intervention. To accomplish this objective, we will utilize a within-subjects multiple baseline design. The children will be randomized to their start times. Clinical ratings, as well as parent- and child- report ratings will be obtained every two weeks (plus or minus seven days) during both the baseline and active periods. This is not an RCT. All children will receive active CBT following variable (randomized) start times. Consistent with the manual we will continue to meet with children and their parents utilizing newly manualized exposure-based CBT procedures, such as eliciting hierarchies of irritability inducing events, exposure exercises (e.g., in-vivo, role-play, imaginal) and parent training. We will conduct the CBT on N=40 youth with severe, impairing irritability. Primary outcome measures for CBT will assess changes in irritability using the ARI (clinician-rated, parent-rated, and child-rated) and CGI-I.

Secondary Objective 1a and 1b: Assess the effect of IBT on clinical measures of depression, anxiety, and functional impairment.

Secondary Objective 2: Assess the effect of the CBT for irritability on clinical measures of depression, anxiety, and functional impairment.

Subjects can participate in one or both of these potential treatments. If they opt to do both, there will be a four-week wash-out period between treatments.

STUDY POPULATION:

The study is taking place at the National Institutes of Health (NIH). All outpatients, ages 8-17, enrolled in NIMH-DIRP Protocol 02-M-0021, who are in stable treatment in the community will be invited to participate in this study.

DESIGN:

The first part of the protocol will involve conducting a randomized controlled trial of IBT in 40 youths who meet criteria for DMDD. The goal of this novel, potential treatment is to decrease the severity of the child s irritability.

The second part of the protocol will involve conducting a randomized within-subjects multiple-baseline trial of CBT targeting severe irritability including N=40 youth.

Subjects can elect to participate in the IBT randomized controlled trial only, CBT treatment or both. If subjects elect to participate in both IBT and CBT, there will be a one-month wash-out period in between.

OUTCOME MEASURES:

The main outcome measures will assess changes in irritability using the ARI (clinician-rated, parent-rated, and child-rated, original and revised versions for IBT and CBT, respectively) and CGI-I. Secondary measures include parent and self-report measures of irritability, depression, anxiety, anger, social status, and aggression, as well as clinician ratings of depression, anxiety, and impairment. Data for ecological momentary assessments (EMA) will be collected using secure technology, with procedures approved by the NIMH ISSO; subjects and their caregivers will be asked a set of questions relating to recent experiences and emotions

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria for both Interpretation Bias Training and Cognitive Behavioral Therapy Studies:

1. Age 8-17 years
2. Must be enrolled into NIMH DIRP protocol 02-M-0021, Characterization and Pathophysiology of Severe Mood and Behavioral Dysregulation in children and youth.
3. Must meet DSM 5 diagnostic criteria for DMDD which are (for CBT, must meet lifetime history of either DMDD or one of two core DMDD criteria [b or c]):

   * Must meet all of the following:

     1. Diagnosis must first be made between ages 6-18 years
     2. Abnormal mood (specifically, anger and/or irritability), present at least half of the day most days, and of sufficient severity to be noticeable by people in the child s environment (e.g. parents, teachers, peers).
     3. Compared to his/her peers, the child exhibits markedly increased reactivity to negative emotional stimuli that is manifest verbally or behaviorally. For example, the child responds to frustration with extended temper tantrums (inappropriate for age and/or precipitating event), verbal rages, and/or aggression toward people or property. Such events occur, on average, at least three times a week.
   * The symptoms in b and c above are currently present and have been present for at least 12 months without any symptom-free periods exceeding two months.
   * The onset of symptoms must be prior to age 10 years.
   * The symptoms are severe in at least one setting (e.g. violent outbursts, assaultiveness at home, school, or with peers). In addition, there are at least mild symptoms (verbal aggression) in a second setting.
4. Patients must be fluent in English

   1. All instruments have not been validated in other languages.
   2. Psychotherapy will be designed and conducted in English.
5. On the basis of record review and interviews with child and parent, the research team agrees that the child s response to his/her current treatment is no more than minimal (i.e. CGI-S of 3 or more).
6. Must have no planned changes in outpatient psychiatric treatment regimen, which can include psychotropic medications and/or psychotherapeutic interventions, two weeks prior to enrollment and throughout the three weeks of training and post-training assessment.

EXCLUSION CRITERIA:

Exclusion criteria both Interpretation Bias Training and Cognitive Behavioral Therapy Studies:

1. The individual exhibits any of these cardinal bipolar symptoms:

   1. Elevated or expansive mood.
   2. Grandiosity or inflated self-esteem.
   3. Decreased need for sleep.
   4. Increase in goal-directed activity (this can result in the excessive involvement in pleasurable activities that have a high potential for painful consequences).
   5. A history of hypomanic or manic symptoms that occurred in distinct episodes lasting more than 1 day.
2. Meets DSM 5 criteria for schizophrenia, schizophreniform disorder, schizoaffective illness, Autism Spectrum Disorder, or posttraumatic stress disorder.
3. IQ<70
4. The symptoms are due to the direct physiologic effects of a drug of abuse, or to a general medical or neurological condition.
5. Meets criteria for alcohol or substance abuse three months prior to enrollment.
6. Meets DSM 5 criteria for current major depressive disorder. The rationale for the exclusion of youth with MDD is because the two novel interventions being tested are contraindicated for those with major depressive disorder. However, there is no contraindication to participation for those with treated/resolved or remitted major depressive disorder; only those with a current diagnosis need to be excluded.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All outpatients, ages 8-17, enrolled in NIMH-DIRP Protocol 02-M-0021, and who are on stable, community treatment will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-11-17 (Actual); Primary Completion 2028-05-08 (Estimated); Study Completion 2028-05-08 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression--Improvement score | Every two weeks
  Clinician administered measure to assess clinical symptoms
Affective Reactivity Index (ARI) | Every two weeks
  Clinician administered measure to assess clinical symptoms

SECONDARY OUTCOMES:
parent and self-report measures of irritability, depression, anxiety, anger, social status, and aggression, as well as clinician ratings of depression, anxiety, and impairment | Weekly
  Self- and parent-report measures to assess clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Brotman, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared.

REFERENCES:
- [Background] Leibenluft E. Severe mood dysregulation, irritability, and the diagnostic boundaries of bipolar disorder in youths. Am J Psychiatry. 2011 Feb;168(2):129-42. doi: 10.1176/appi.ajp.2010.10050766. Epub 2010 Dec 1. PMID 21123313
- [Background] Leibenluft E, Stoddard J. The developmental psychopathology of irritability. Dev Psychopathol. 2013 Nov;25(4 Pt 2):1473-87. doi: 10.1017/S0954579413000722. PMID 24342851
- [Background] Brotman MA, Kircanski K, Stringaris A, Pine DS, Leibenluft E. Irritability in Youths: A Translational Model. Am J Psychiatry. 2017 Jun 1;174(6):520-532. doi: 10.1176/appi.ajp.2016.16070839. Epub 2017 Jan 20. PMID 28103715
- [Derived] Naim R, German RE, White J, Pandya U, Dombek K, Clayton M, Perlstein S, Henry LM, Kircanski K, Lorenzo-Luaces L, Brotman MA. Treatment adherence, therapeutic alliance, and clinical outcomes during an exposure-based cognitive-behavioral therapy for pediatric irritability. BMC Psychiatry. 2025 Feb 26;25(1):181. doi: 10.1186/s12888-025-06601-0. PMID 40012036
- [Derived] Grasser LR, Erjo T, Goodwin MS, Naim R, German RE, White J, Cullins L, Tseng WL, Stoddard J, Brotman MA. Can peripheral psychophysiological markers predict response to exposure-based cognitive behavioral therapy in youth with severely impairing irritability? A study protocol. BMC Psychiatry. 2023 Dec 11;23(1):926. doi: 10.1186/s12888-023-05421-4. PMID 38082431
- [Derived] Linke JO, Haller SP, Xu EP, Nguyen LT, Chue AE, Botz-Zapp C, Revzina O, Perlstein S, Ross AJ, Tseng WL, Shaw P, Brotman MA, Pine DS, Gotts SJ, Leibenluft E, Kircanski K. Persistent Frustration-Induced Reconfigurations of Brain Networks Predict Individual Differences in Irritability. J Am Acad Child Adolesc Psychiatry. 2023 Jun;62(6):684-695. doi: 10.1016/j.jaac.2022.11.009. Epub 2022 Dec 21. PMID 36563874
- [Derived] Haller SP, Archer C, Jeong A, Jaffe A, Jones EL, Harrewijn A, Naim R, Linke JO, Stoddard J, Brotman MA. Changes in Internalizing Symptoms During the COVID-19 Pandemic in a Transdiagnostic Sample of Youth: Exploring Mediators and Predictors. Child Psychiatry Hum Dev. 2024 Feb;55(1):206-218. doi: 10.1007/s10578-022-01382-z. Epub 2022 Jul 6. PMID 35794298
- [Derived] Haller SP, Stoddard J, Botz-Zapp C, Clayton M, MacGillivray C, Perhamus G, Stiles K, Kircanski K, Penton-Voak IS, Bar-Haim Y, Munafo M, Towbin KE, Brotman MA. A Randomized Controlled Trial of Computerized Interpretation Bias Training for Disruptive Mood Dysregulation Disorder: A Fast-Fail Study. J Am Acad Child Adolesc Psychiatry. 2022 Jan;61(1):37-45. doi: 10.1016/j.jaac.2021.05.022. Epub 2021 Jun 17. PMID 34147585
- [Derived] Naim R, Kircanski K, Gold A, German RE, Davis M, Perlstein S, Clayton M, Revzina O, Brotman MA. Across-subjects multiple baseline trial of exposure-based cognitive-behavioral therapy for severe irritability: a study protocol. BMJ Open. 2021 Mar 10;11(3):e039169. doi: 10.1136/bmjopen-2020-039169. PMID 33692176
- [Derived] Linke JO, Abend R, Kircanski K, Clayton M, Stavish C, Benson BE, Brotman MA, Renaud O, Smith SM, Nichols TE, Leibenluft E, Winkler AM, Pine DS. Shared and Anxiety-Specific Pediatric Psychopathology Dimensions Manifest Distributed Neural Correlates. Biol Psychiatry. 2021 Mar 15;89(6):579-587. doi: 10.1016/j.biopsych.2020.10.018. Epub 2020 Nov 9. PMID 33386133
- [Derived] Linke J, Kircanski K, Brooks J, Perhamus G, Gold AL, Brotman MA. Exposure-Based Cognitive-Behavioral Therapy for Disruptive Mood Dysregulation Disorder: An Evidence-Based Case Study. Behav Ther. 2020 Mar;51(2):320-333. doi: 10.1016/j.beth.2019.05.007. Epub 2019 May 21. PMID 32138941
- [Derived] Haller SP, Kircanski K, Stringaris A, Clayton M, Bui H, Agorsor C, Cardenas SI, Towbin KE, Pine DS, Leibenluft E, Brotman MA. The Clinician Affective Reactivity Index: Validity and Reliability of a Clinician-Rated Assessment of Irritability. Behav Ther. 2020 Mar;51(2):283-293. doi: 10.1016/j.beth.2019.10.005. Epub 2019 Nov 27. PMID 32138938
- [Derived] Cardinale EM, Kircanski K, Brooks J, Gold AL, Towbin KE, Pine DS, Leibenluft E, Brotman MA. Parsing neurodevelopmental features of irritability and anxiety: Replication and validation of a latent variable approach. Dev Psychopathol. 2019 Aug;31(3):917-929. doi: 10.1017/S095457941900035X. Epub 2019 May 8. PMID 31064595
- [Derived] Haller SP, Stoddard J, MacGillivray C, Stiles K, Perhamus G, Penton-Voak IS, Bar-Haim Y, Munafo MR, Brotman MA. A double-blind, randomized, placebo-controlled trial of a computer-based Interpretation Bias Training for youth with severe irritability: a study protocol. Trials. 2018 Nov 14;19(1):626. doi: 10.1186/s13063-018-2960-5. PMID 30428909
- [Derived] Stringaris A, Vidal-Ribas P, Brotman MA, Leibenluft E. Practitioner Review: Definition, recognition, and treatment challenges of irritability in young people. J Child Psychol Psychiatry. 2018 Jul;59(7):721-739. doi: 10.1111/jcpp.12823. Epub 2017 Oct 30. PMID 29083031
- [Derived] Brotman MA, Kircanski K, Leibenluft E. Irritability in Children and Adolescents. Annu Rev Clin Psychol. 2017 May 8;13:317-341. doi: 10.1146/annurev-clinpsy-032816-044941. PMID 28482689
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-M-0182.html